CLINICAL TRIAL: NCT06793670
Title: The Use of Landiolol in Mitral Valve sUrgery: a raNdomized, Controlled, Double-blind triAl (LUNA)
Brief Title: Landiolol in Mitral Valve Surgery
Acronym: LUNA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PNRR-MCNT2-2023-12377946
Record Dates: First submitted 2025-01-15; First posted 2025-01-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Failure; Low Cardiac Output Syndrome
MeSH Terms: conditions — Heart Failure; Cardiac Output, Low | interventions — landiolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Landiolol (Experimental): intraoperative landiolol, first as low-dose continuous infusion (5 mcg/kg/min) until aortic cross clamping, followed by an intravenous bolus (0.3 mg/kg) after aortic cannulation (but still before aortic cross-clamping) and a further intravenous bolus dose of 0.3 mg/kg as cardioplegia adjuvant added to the first administered cardioplegic solution.
  Interventions: Drug: Landiolol
- Placebo (Placebo Comparator): intraoperative equivolume placebo normal saline solution, first as low-dose continuous infusion until aortic cross clamping, followed by an intravenous bolus after aortic cannulation and a further equivolume quantity added to the first administered cardioplegic solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Landiolol — Intravenous infusion of landiolol
  Arms: Landiolol
Drug: Placebo — Intravenous infusion of saline solution of NaCl 0.9%
  Arms: Placebo

SUMMARY:
Chronic mitral regurgitation is the most common valvular abnormality worldwide, it occurs in 10% of the general population and its prevalence increases with age. When left untreated, it can lead to left ventricular dysfunction and cause disabling symptoms (e.g., fatigue and dyspnea), life-threatening complications (e.g., ventricular dilation, congestive heart failure) and death. Surgical correction of chronic mitral regurgitation before irreversible changes happen can be curative. Open surgical valve repair or replacement are accomplished through cardiopulmonary bypass and cardioplegic arrest. Myocardial protection is essential to guarantee an uneventful perioperative course since a not-well protected heart may lead to postoperative low-cardiac output syndrome. This occurs in 30% of high-risk patients who undergo elective cardiac surgery and is associated with 20% mortality. Cardioplegia preserves the heart during ischemic arrest by reducing its metabolic demand. The most effective cardioplegia for protection in adult cardiac surgery remains unknown and improving the protection of the heart during the ischemic arrest may potentially improve patients' postoperative outcomes. Pharmacological adjuvants to the cardioplegic solutions have been tested to mitigate the ischaemic-reperfusion injury following cardiac surgery. Ultra-short acting beta-blockers (e.g., esmolol, landiolol) decrease intraoperative myocardial metabolic demand and suppress the sympathetic response to surgical stimuli while exhibiting limited adverse effects. Few studies with limited sample size investigated the role of ultra-short acting beta-blockers in reducing perioperative ischaemia and arrhythmia after cardiac surgery. When ultra-short acting beta-blockers were administered before aortic cross-clamping and as cardioplegia adjuvant we observed a trend towards a reduction in postoperative low-cardiac output syndrome (13/98 vs 6/102; p=0.08) and in the rate of hospital re-admission at one year (26/95 v 16/96, p=0.08) with an increase in the number of patients with ejection fraction >60% at hospital discharge (4/95 vs 11/92, p=0.06) (Zangrillo 2021). However, despite a growing body of literature exploring the role of ultra-short acting beta-blockers in enhancing myocardial protection during on-pump cardiac surgery, further high-quality evidence is needed before this practice can be established as standard routine care. Hence, we designed a randomized, placebo-controlled trial involving 1500 patients undergoing open mitral valve surgery to assess the effect of administering landiolol as cardioplegia adjuvant to reduce the occurrence of postoperative low-cardiac output syndrome. Successful results would have a significant impact on short and long-term complications.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years;
* Elective mitral valve repair or replacement surgery with planned cardiopulmonary bypass via midline sternotomy or minithoracotomy;
* Preoperative evidence of left ventricular end-systolic diameter >40 mm and/or left ventricular end-diastolic diameter >60 mm and/or left ventricular ejection fraction<60%;
* Signed informed consent.

Exclusion Criteria:

* Need for preoperative dialysis;
* Hepatic dysfunction (defined as Child-Pugh class C);
* History of previous unusual response to beta-blockers;
* Urgent or emergency surgery;
* Patient already in need of mechanical circulatory support before surgery (except for IABP);
* Pregnancy as documented by a pregnancy test performed in the last 72h before surgery;
* Patients with preoperative evidence of hypernatremia (serum sodium concentration: > 160 mmol/L);
* Patients with preoperative evidence of hyperchloremia (serum chloride concentration: >115 mmol/L);
* Patients with hypersensitivity to the active substance or to any of the excipients;
* Patients with severe bradycardia (less than 50 beats per minute) sick sinus syndrome, severe atrioventricular nodal conductance disorders or 2nd -3rd degree atrioventricular block and without a pacemaker;
* Patients with cardiogenic shock, severe hypotension (MAP<50 mmHg), decompensated heart failure or severe pulmonary hypertension (PAPs >70 mmHg);
* Patients with non-treated phaeochromocytoma;
* Patients with acute asthmatic attack;
* Patients with severe, uncorrectable metabolic acidosis.
* Participation in a clinical trial in which an investigational drug was administered within 30 days of screening or within the 5 half-lives of the study drug, whichever is longer.
* Planned use of ultra-short acting beta-blockers as intraoperative cardiac protective strategy.
* Refusal or inability to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of the occurrence of postoperative low-cardiac output syndrome (LCOS) | Until ICU discharge, an average of 4 days
  The primary outcome will be the reduction of the occurrence of postoperative low-cardiac output syndrome, defined following Cholley et al. 2017 JAMA as the presence of at least one of the following:
  1. need of prolonged catecholamine infusion (persisting beyond 48 hours after the initiation of the study drug);
  2. need of circulatory mechanical assist devices in the postoperative period (if an intra-aortic balloon pump was inserted preventively, the criteria will be met if patients are not weaned from the balloon within 96 hours);
  3. need for renal replacement therapy at any time during the intensive care unit stay.

SECONDARY OUTCOMES:
Patients requiring prolonged (>48 h) catecholamine infusion | Until ICU discharge, an average of 4 days
Patients with increased postoperative cardiac biomarkers (Troponin I or T) | Up to 48 hours.
Patients with a reduction in left ventricular ejection fraction | Until hospital discharge, an average of 10 days
Number of patients readmitted to hospital for cardiac reasons | 1 year
EQ-5D-5L questionnaire | 1 year
Death | 1 year

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Ospedale Cesare Arrigo, Alessandria, Piedmont
  - A. O. Ordine Mauriziano di Torino, Torino, TO
  - AOU di Alessandria, Alessandria
  - Azienda Ospedaliero Universitaria Policlinico "G.Rodolico - San Marco", Catania
  - AOU Careggi, Florence
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - IRCCS San Martino di Genova, Genova
  - Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - AOR San Carlo, Potenza
  - Maria Cecilia Hospital S.p.A., Ravenna

IPD SHARING:
Plan to Share IPD: No